CLINICAL TRIAL: NCT02440308
Title: 68Ga-DOTA-Bombesin PET/MRI in the Evaluation of Patients With Prostate Cancer: A Feasibility Study
Brief Title: 68Ga-DOTA-Bombesin PET/MRI in Imaging Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-32319; PROS0069 (Other: OnCore); NCI-2015-00673 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA124435 (NIH)
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — BAY 86-7548; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (1):
- 68Ga-DOTA-Bombesin PET/MRI (Experimental): Patients receive 68Ga-DOTA-Bombesin IV and then undergo PET/MRI approximately 1 hour later.
  Interventions: Drug: 68Ga-DOTA-Bombesin; Procedure: Magnetic Resonance Imaging (MRI) scan; Procedure: Positron Emission Tomography (PET) scan

INTERVENTIONS:
Drug: 68Ga-DOTA-Bombesin — 68Ga-DOTA-Bombesin is a gallium-68-labeled gastrin-releasing peptide receptor (GRPr) antagonist. DOTA is [4,7,10-Tris-(carboxymethyl)-1,4,7,10-tetraazacyclododec-1-yl]-acetyl.
  68Ga-DOTA-Bombesin is administered intravenously (IV)
  Other Names: 68Ga-DOTA RM2; BAY 86-7548; Gallium-68-labeled GRPr Antagonist
Procedure: Magnetic Resonance Imaging (MRI) scan
  Other Names: Nuclear Magnetic Resonance (NMR) scan
Procedure: Positron Emission Tomography (PET) scan
  Other Names: Proton magnetic resonance spectroscopic imaging

SUMMARY:
This clinical trial studies the use of gallium-68 (68Ga)-DOTA-Bombesin as the imaging agent for positron emission tomography (PET)/magnetic resonance imaging (MRI), collectively PET-MRI, in patients with prostate cancer. PET uses a radioactive substance called 68Ga-DOTA-Bombesin, which attaches to tumor cells with specific receptors on their surfaces. The PET scanner takes pictures that capture where the radioactive drug is "lighting up" and attaching to tumor cells, which may help doctors recognize differences between tumor and healthy prostate tissue. MRI uses radio waves and a magnet to make a picture of areas inside the body. Using 68Ga-DOTA-Bombesin in diagnostic procedures, such as PET/MRI, may allow doctors to identify smaller tumors than standard imaging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility and biodistribution of 68Ga-DOTA-Bombesin (BAY 86-7548 or 68Ga-DOTA RM2).

OUTLINE:

Patients receive 68Ga-DOTA-Bombesin intravenously (IV) and then undergo PET/MRI approximately 1 hour later.

After completion of study, patients are followed up at 24 hours and 1 week.

ELIGIBILITY:
INCLUSION CRITERIA

* Provides written informed consent
* Known diagnosis of prostate cancer
* Patient has suspected recurrence based on biochemical data [prostate-specific antigen (PSA) > 2 ng/mL]
* Able to remain still for duration of each imaging procedure (about one hour)

EXCLUSION CRITERIA

* Unable to provide informed consent
* Inability to lie still for the entire imaging time
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance
* Metallic implants

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

REFERENCES:
- [Derived] Minamimoto R, Hancock S, Schneider B, Chin FT, Jamali M, Loening A, Vasanawala S, Gambhir SS, Iagaru A. Pilot Comparison of (6)(8)Ga-RM2 PET and (6)(8)Ga-PSMA-11 PET in Patients with Biochemically Recurrent Prostate Cancer. J Nucl Med. 2016 Apr;57(4):557-62. doi: 10.2967/jnumed.115.168393. Epub 2015 Dec 10. PMID 26659347

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 68Ga-DOTA-Bombesin PET/MRI
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 68Ga-DOTA-Bombesin PET/MRI
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 73.3 [60.8 to 83.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Normal Biodistribution of 68Ga-DOTA-Bombesin
Description: Radiopharmaceutical uptake in normal organs will be evaluated visually and measured semi-quantitatively using standardized uptake values (SUV) derived from the PET/CT scan software in patients with prostate cancer. Uptake values in different tissues will be measured as SUVmean (mean value for SUV). SUVmean values reflect relative uptake of the radiolabel into the tissue.
Time Frame: 1 hour
Population: All participants were averaged to provide SUVmean uptake in normal organs.
Measure: Mean (Standard Deviation); unit: SUV-mean
Arm/Group | 68Ga-DOTA-Bombesin PET/MRI
Number analyzed (Participants) | 10
SUV-mean
  Ascending aorta (blood pool) | 2.28 (0.68)
  Bladder | 121.55 (67.45)
  Brain cortex (frontal lobe) | 0.08 (0.04)
  Cerebellum | 0.10 (0.05)
  Cervical vertebrae | 0.70 (0.19)
  Choroid plexus | 0.25 (0.16)
  Colon | 2.01 (0.74)
  Esophagus | 4.08 (1.51)
  Extra focal uptakes | 12.72 (7.77)
  Femur | 0.34 (0.12)
  Liver | 1.94 (0.48)
  Lung | 0.48 (0.16)
  Gluteal fat | 0.60 (0.19)
  Gluteal muscle | 0.79 (0.41)
  Humerus | 0.53 (0.17)
  Kidney | 9.51 (6.15)
  Lumbar vertebrae | 0.75 (0.28)
  Pancreas | 52.02 (16.74)
  Parotid gland | 0.99 (0.23)
  Sacrum | 0.69 (0.36)
  Spleen | 1.62 (0.49)
  Small bowel | 2.40 (0.57)
  Stomach | 2.48 (0.73)
  Submandibular gland | 1.18 (0.45)
  Thoracic vertebrae | 0.91 (0.32)
  Thyroid | 1.31 (0.29)

2. Secondary Outcome: 68Ga-DOTA-Bombesin Feasibility
Description: Feasibility of 68Ga-DOTA-Bombesin as a radiopharmaceutical for PET/MRI was assessed as the percentage of enrolled subjects who complete the examination, and for which the PET/MRI data were evaluable.
Time Frame: Up to 1 week
Population: Includes all participants enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | 68Ga-DOTA-Bombesin PET/MRI
Number analyzed (Participants) | 10
percentage of participants | 100

ADVERSE EVENTS:
Arm/Group | 68Ga-DOTA-Bombesin PET/MRI
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes